CLINICAL TRIAL: NCT02241304
Title: Neurostimulation and Electromyographic Assessment of the TetraGraph (NEAT) In Patients (NEAT-3)
Acronym: NEAT-3
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, MD, PHD, University of Debrecen
Other Study IDs: ADBV-ABS-0214-NEAT-3H; 028605/2014/OTIG (Registry Identifier: The Office for Health Authorization and Administrative Procedures (EEKH)); DE RKEB/IKEB 4170-2014 (Registry Identifier: Regional and Institutional Ethics Committee, Medical and Health Science Center, University of Debrecen)
Record Dates: First submitted 2014-07-08; First posted 2014-09-16 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Neuromuscular Blockade
Keywords: electromyography; neuromuscular blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elective surgery with muscle relaxation: ASA I-II-III patients. Fentanyl (2-3 ug/kg) - Propofol (2 mg/kg) induction, sevoflurane anesthesia, type and dose of muscle relaxant up to the decision of attending anesthetist. Neuromuscular stimulation with TetraGraph (30mA current intensity, 0.2 msce pulse duration, 20 sec intervals)

SUMMARY:
TetraGraph is a newly developed EMG-based, quantitative, battery-powered neuromuscular monitoring system intended for daily clinical use. The primary aim of this clinical investigation is to examine the applicability (ease of use, equipment need, etc.), repeatability (precision or internal consistency) and performance (signal quality, accuracy of outcome, voltage of stimulation output before and during a stimulus) of the Tetragraph device in patients undergoing elective surgeries requiring neuromuscular blockade.

DETAILED DESCRIPTION:
The TetraGraph will be tested in 50 consenting patients undergiong elective surgeries requiring neuromuscular blockade. The left of right hand of the patients will be randomly studied. After the induction of anesthesia but before the administration of muscle relaxant train-of-four (TOF) stimulation will be started with 30 mA current intensity, 0.2 msec pulse duration at 20 sec intervals. The stimulation will be left to run until extubation. The TetraGraph device will be set not to show measurement results on the screen but save them on the SD card for later analysis. This way TetraGraph will not influence clinical decisions and patient care. During the operations we will record the number of muscle twitches in return to stimulation, the time and dose of muscle relaxant and opioid administration, the time of use of electrocautery and the skin temperature.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. American Society of Anesthesiology (ASA) physical status I-III criteria (Table I).
3. Subject has provided written informed consent.

Exclusion Criteria:

1. Presence of an underlying neuromuscular disease.
2. Presence of renal or hepatic disease.
3. Subject has open skin sores in the locations needed for electrode application (forearms).
4. Patient is taking anti-seizure medication
5. Patient is taking oral anti-cholinesterase (e.g., therapy for myasthenia gravis)
6. Magnesium sulfate administration is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgeries requiring muscle relaxation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary performance assessment of TetraGraph device | participants will be followed for the duration of their hospital stay, an expected avarage of five days
  The primary objective of this study is to provide safety & performance data of the TetraGraph device in anesthetized patients. Performance will be assessed post hoc by analyzing objective EMG data from the SD card and correlating the responses to annotations made during the surgical procedure (e.g., correlating the EMG responses to the time of NMBA or reversal agent administration). No clinical decisions will be made based on any objective measurements made by the TetraGraph. There are no specific timepoints concerning the primary outcome measure of the study.

SECONDARY OUTCOMES:
Secondary performance assessment of TetraGraph Device | participants will be followed for the duration of the hospital stay, an expected avarage of 5 days
  The secondary outcome measures is a composite of several safety and performance data examined during the operations and the hospital stay:
  1. Acceptable levels of electrical noise when no stimulus is being applied;
  2. Ensuring that the stimulus artifact does not obscure the EMG response when a stimulus is applied;
  3. Appearance of an EMG response at threshold stimulation levels, just sufficient to elicit a palpable twitch response;
  4. Consistency of the EMG response amplitudes during repeated (ST and TOF) protocols (variability <10%);
  5. Consistency of EMG response characteristics independent of patient age, gender, or weight;
  6. Consistency of EMG response characteristics independent whether the right or left arm is stimulated;
  7. Skin reaction to stimulation or recording electrodes;
  8. Overall usability of the device for clinicians and operators; collecting recommendations for improving ease of use.
Safety of TetraGraph device | participants will be followed for the duration of hospital stay, an expected avarage of 5 days
  The safety of Tetragraph device will be assesses by checking the stimulating and recording electrode positions for skin reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Bela Fulesdi, MD,PhD,DSci, Principal Investigator — UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care Debrecen, Hungary, 4032
Locations (1):
- University of Debrecen, Debrecen, Hungary

REFERENCES:
- [Background] 1. Gätke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Acta Anaesthesiol Scand 2002;46:207-13. 2. Berg H, Viby-Mogensen J, Roed J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Acta Anaesthesiol Scand 1997;41:1095-103. 3. Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Anesth Analg 2008;107:130-7. 4. Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Nisman M. Anesthesiology 2008;109:389-98. 5. Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Vender JS, Gray J, Landry E, Gupta DK. Anesthesiology 2011;115:946-54. 6. Murphy GS, Brull SJ. Anesth Analg 2010;111:120-8. 7. Hemmerling TM, Le N. Can J Anesth 2007;54: 58-72. 8. Gätke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Acta Anaesthesiol Scand 2002; 46: 207-13. 9. Brull SJ, Silverman DG. Anesth Analg 1993;77:352-5. 10. Grayling M, Sweeney BP. Anaesthesia 2007; 62:806-9. 11. Liang SS, Stewart PA, Phillips S. Anesth Analg 2013;117:373-9.